CLINICAL TRIAL: NCT02508207
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Exploratory Study to Evaluate Effects of VX-661 in Combination With Ivacaftor on Lung and Extrapulmonary Systems in Subjects Aged 18 Years and Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: A Phase 2 Study to Evaluate Effects of VX-661/Ivacaftor on Lung and Extrapulmonary Systems in Subjects With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX14-661-111
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor; tezacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to tezacaftor (TEZ)/ivacaftor (IVA) fixed dose combination (FDC) tablet orally once daily in the morning followed by placebo matched to IVA tablet orally once daily in the evening for 29 days.
  Interventions: Drug: Tezacaftor/Ivacaftor matching placebo; Drug: Ivacaftor matching placebo
- TEZ/IVA (Experimental): Participants received 100 milligram (mg) TEZ/150 mg IVA FDC tablet orally once daily in the morning followed by 150 mg IVA tablet orally once daily in the evening for 29 days.
  Interventions: Drug: Tezacaftor/Ivacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Tezacaftor/Ivacaftor — Tezacaftor/Ivacaftor FDC
  Arms: TEZ/IVA
Drug: Ivacaftor
  Arms: TEZ/IVA
Drug: Tezacaftor/Ivacaftor matching placebo
  Arms: Placebo
Drug: Ivacaftor matching placebo
  Arms: Placebo

SUMMARY:
To evaluate the clinical mechanisms of action in lung and extrapulmonary systems of VX-661 (tezacaftor; TEZ) in combination with ivacaftor (IVA) (TEZ/IVA) in participants with cystic fibrosis (CF) who are homozygous for the F508del mutation on the CF transmembrane conductance regulator (CFTR) gene.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, homozygous for the F508del CFTR mutation
* Confirmed diagnosis of CF by sweat chloride testing
* Forced Expiratory Volume in 1 Second (FEV1) ≥40% and ≤90% of predicted normal for age, sex, and height at Screening Visit
* Stable CF disease as judged by the investigator.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before Day 1
* History or evidence of clinically significant findings on ophthalmologic examination during the Screening Period.
* History of solid organ or hematological transplantation
* Pregnant or nursing females
* Participants who have had radiation exposure within 1 year before the first mucociliary clearance (MCC) procedure that would cause them to exceed federal regulations by participating in this study
* In the opinion of the investigator, unable to adequately perform inhalation maneuvers during the MCC procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Birmingham, Alabama
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | TEZ/IVA
Started | 7 | 27
Completed | 7 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo matched to TEZ/IVA FDC tablet orally once daily in the morning followed by placebo matched to IVA tablet orally once daily in the evening for 29 days.
- TEZ/IVA: Participants received 100 mg TEZ/150 mg IVA FDC tablet orally once daily in the morning followed by 150 mg IVA tablet orally once daily in the evening for 29 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | TEZ/IVA | Total
Number analyzed (Participants) | 7 | 27 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (11.8) | 32.1 (8.6) | 33.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 15 | 19
  Male | 3 | 12 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 27 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 27 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mucociliary Clearance (MCC): Percentage of Whole-lung Clearance [Mean (Standard Deviation); unit: percentage of whole-lung clearance] — MCC was assessed using an imaging technique that enables the tracking of mucus within the airways. MCC was expressed as the percentage of whole-lung clearance through 60 minutes at Baseline.
  percentage of whole-lung clearance | 15.3 (15.1) | 18.4 (11.3) | 17.8 (12.0)
Small-bowel Area Under the Curve (AUC) Over 1-minute Mean pH Increments [Mean (Standard Deviation); unit: pH minutes] — Small-bowel AUC through 30 minutes of 1 minute mean pH profile through gastric emptying at Baseline was reported.
  pH minutes | 5.8 (0.4) | 5.7 (0.6) | 5.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Mucociliary Clearance (MCC) at Day 28
Description: MCC was assessed using an imaging technique that enables the tracking of mucus within the airways. MCC was expressed as the percentage of whole-lung clearance through 60 minutes at Baseline and Day 28.
Time Frame: Baseline, Day 28
Population: The Full Analysis Set (FAS) included all randomized participants who carry the relevant cystic fibrosis transmembrane conductance regulator (CFTR) allele and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of whole-lung clearance
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 7 | 27
percentage of whole-lung clearance | -0.5 (11.2) | -0.9 (12.1)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p = 0.7151, t-test, 2 sided — p-value for within TEZ/IVA group was analyzed using a 2-sided, paired, t-test at a 5% level of significance

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 28
Description: Percent predicted FEV1 is the ratio of FEV1 to the predicted FEV1, expressed as a percentage. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 28
Population: The FAS was used.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 7 | 27
percentage of predicted FEV1 | -0.4 (5.9) | 2.4 (3.1)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p = 0.0004, t-test, 2 sided — p-value for within TEZ/IVA group was analyzed using a 2-sided, paired, t-test at a 5% level of significance

3. Secondary Outcome: Absolute Change From Baseline in Small-bowel Area Under the Curve (AUC) Over 1-minute Mean pH Increments at Day 29
Description: Absolute change from Baseline in small bowel AUC over 1-minute mean pH increments through 30 minutes at Day 29 was assessed.
Time Frame: Baseline, Day 29
Population: The FAS was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pH minutes
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 6 | 23
pH minutes | 0.3 (0.5) | -0.2 (0.8)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p = 0.3345, t-test, 2 sided; p-value for within TEZ/IVA group was analyzed using a 2-sided, paired, t-test at a 5% level of significance

4. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride at Day 29
Time Frame: Baseline, Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 7 | 23
millimoles per liter | -0.2 (6.0) | -8.4 (9.2)
Statistical Analysis 1: Comparison: TEZ/IVA; Test type: Other; p = 0.0002, t-test, 2 sided — p-value for within TEZ/IVA group was analyzed using a 2-sided, paired, t-test at a 5% level of significance

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Day 57
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEZ/IVA
Number analyzed (Participants) | 7 | 27
Participants
  Participants with SAEs | 0 | 0
  Participants with AEs | 2 | 24

ADVERSE EVENTS:
Time Frame: Baseline up to Day 57: 29 days of dosing + 28 days of safety follow up
Description: Other adverse events table reports the participants with adverse events that exceed a frequency threshold of at least 5% within any arm of the study.
Arm/Group | Placebo | TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/27
Other Adverse Events (participants affected / at risk) | 2/7 | 18/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | TEZ/IVA (N=27)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT02508207/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT02508207/SAP_001.pdf